CLINICAL TRIAL: NCT02840240
Title: A Randomized Controlled Trial to Determine the Effect of Gabapentin Enacarbil on Opioid Consumption and Pain Scores in Patients Having Hip and Knee Arthroplasties With Spinal Anesthesia
Brief Title: Effect of Gabapentin Enacarbil on Opioid Consumption and Pain Scores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-479
Record Dates: First submitted 2016-05-23; First posted 2016-07-21 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin enacarbil (Experimental): Patients going through elective hip or knee replacement surgery with spinal anesthesia will receive Gabapentin enacarbil for 5 days
  Interventions: Drug: Gabapentin enacarbil
- Placebo (Placebo Comparator): Patients going through elective hip or knee replacement surgery with spinal anesthesia will receive placebo for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin enacarbil — 600 mg BID 1 day pre-op and 2 hours before surgery, 6 hours after surgery, 600 mg BID 3 days post-operative
  Other Names: Xenoport
  Arms: Gabapentin enacarbil
Drug: Placebo — 600 mg BID taken 1 day pre-op and 2 hours before surgery, 6 hours after surgery, 600 mg 3 days post-operative
  Arms: Placebo

SUMMARY:
Opioids are effective analgesics, but cause side effects including sedation, respiratory depression, low blood pressure, nausea, and constipation. Gabapentin enacarbil, which is a FDA approved drug for post herpetic neuralgia (nerve pain related to shingles) and restless leg syndrome, may decrease your need for narcotics and thus decrease the risk of side effects. The investigator hopes this study will determine if gabapentin enacarbil decreases opioid consumption and pain after surgery.

Patients having elective hip and knee surgery will be asked to participate in the study. Patients will be randomized to Gabapentin enacarbil 600mg twice per day for 5 days or Placebo twice per day for 5 days.

One day prior to surgery the patient will take Gabapentin enacarbil 600mg or placebo 600mg twice a day with meals. On the day of surgery, the patient will take Gabapentin enacarbil 600mg or placebo 600mg two hours before the surgical procedure. Six hours after the completion of surgery, the patient will receive Gabapentin enacarbil 600mg or placebo 600mg. If the patient is sent home, the patient will be given 6 Gabapentin enacarbil 600mg or placebo 600mg pills to take home along with instructions. However, if the patient remains hospitalized, on the first day after the surgery, the patient will have pain assessed in the morning using a numerical rating score. The patient's quality of recovery will be evaluated using a questionnaire and the patient will receive Gabapentin enacarbil 600mg or placebo 600mg twice a day with meals. The second and third day the patient is in the hospital, the patient will have pain assessed in the morning using a numerical rating score and the patient will receive Gabapentin enacarbil 600mg or placebo 600mg twice a day with meals. Then, three months after surgery, the patient will receive a phone call to follow-up with possible pain or discomfort the patient may be feeling.

DETAILED DESCRIPTION:
A randomized controlled trial to determine the effect of gabapentin enacarbil on opioid consumption and pain scores in patients having primary hip or knee replacement surgery with spinal anesthesia.

Screening visit

* Consent will be obtained
* Vital Signs
* Physical evaluation
* Medical History
* Laboratory values and medication checked via Epic
* Pain scores using numerical rating scores (NRS)
* Brief pain inventory (BPI)
* Randomization will be to standard management with GEn or to standard management with placebo. Patients will be given GEn 600 mg bid or placebo 600 mg bid for 1 preoperative day and will receive 600 mg GEn or placebo about 2 hours before surgery and then restarted on GEn or placebo 600 mg within 6 hours of surgery, and then 600 mg bid for three additional days.

  2 days prior to surgery Phone call will be made to remind patients to take GEn 600 mg bid or placebo 600 mg bid

  1 day prior to surgery
* vital signs
* GEn 600 mg bid or placebo 600 mg bid
* monitoring and recording of adverse events

Day of Surgery

* Medical History
* Laboratory values and medication checked via Epic
* Patients will be given GEn 600 mg or placebo single dose with sips of water 2 hours before surgery and then restarted within 6 hours of completion of surgery.
* Vital Signs
* Social history
* Demographic data to be obtained includes height (cm), weight (kg), age (yr), gender, (ASA) physical status, and self-declared ethnicity
* Individual risk for nausea and vomiting will be determined using the Apfel score.
* Monitoring and recording of adverse events
* Pain scores using numerical rating scores (NRS) during the PACU stay every 15 minutes for the first hour after surgery

POD 1

* GEn 600 mg bid or placebo 600 mg bid
* Vital Signs
* Monitoring and Recording of adverse events
* Pain scores using numerical rating scores (NRS) in the morning
* Myles QoR scale to formally evaluate quality of recovery

POD 2

* GEn 600 mg bid or placebo 600 mg bid
* Vital Signs
* Monitoring and Recording of adverse events
* Pain scores using numerical rating scores (NRS) in the morning

POD 3

* GEn 600 mg bid or placebo 600 mg bid
* Vital Signs
* Monitoring and Recording of adverse events
* Pain scores using numerical rating scores (NRS) in the morning

  3 Months after surgery
* Phone call will be made to check for any adverse event and with the intention to assess chronic pain.
* Monitoring and recording of adverse events
* Data obtained from electronic medical records will include: operation time, surgery type, intraoperative opioid consumption, postoperative opioid consumption in PACU and in ward, breakthrough pain medication requirements, pain scores in PACU and ward, requirement of antiemetics for nausea and vomiting, requirement of antihistaminic medications, requirement of laxatives for constipation, ambulation time, flatus, ileus, bowel movements, length of stay and any side effects or complications. Preoperative and postoperative laboratory data including but not limited to renal function will also be collected from electronic medical records. Patient functionality will also be recorded including, bathing, toileting, walking and moving.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18-85 years of age.
2. Scheduled for elective knee or hip arthroplasty with spinal anesthesia.

Exclusion Criteria:

1. Creatinine >1.50 mg/dl.
2. History of clinically important current depression or currently on any prescribed anti-depressant medication.
3. Previously enrolled in any Xenoport trial.
4. Use of gabapentin or gabapentinoids (Lyrica, Horizant, Neurontin or Gralise) within one month.
5. Allergy to gabapentin or gabapentinoids (Lyrica, Horizant, Neurontin or Gralise).
6. Women who are pregnant or breastfeeding.
7. History of seizure disorder within the last one-year or taking medications for seizures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin Enacarbil | Placebo
Started | 56 | 51
Completed | 28 | 32
Not Completed | 28 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin Enacarbil | Placebo | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 66 (9) | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 11 | 15 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/white | 25 | 29 | 54
  African American | 2 | 2 | 4
  Other | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: cm] | 169 (11) | 169 (10) | 169 (10)
Weight [Mean (Standard Deviation); unit: kg] | 90 (26) | 90 (20) | 90 (23)

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Average Pain Score in Numerical Rating Scores
Description: Multiple pain measurements (numeric rating scale ranges from 0 to 10, where 0 - no pain and 10 - worse imaginable pain) over 72 hours after the surgery will be summarized by computing time weighted average pain score for each patient
Time Frame: Initial 72 hours after surgery or until discharge, whatever comes first.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin Enacarbil | Placebo
Number analyzed (Participants) | 28 | 32
score on a scale | 4.0 (1.6) | 4.1 (1.7)
Statistical Analysis 1: Comparison: Gabapentin Enacarbil vs Placebo; Test type: Non-Inferiority — Noninferiority deltas were defined a priori as 1.1 for the ratio in geometric means of opioid consumption converted to IV morphine equivalents (ie, no more than 10% difference between group's median doses) and 1 point for pain score (ie, no more than 1 point worse); p = 0.003, Regression, Linear; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.07 to 0.69]

2. Primary Outcome: Cumulative Postoperative Opioid Consumption
Description: The total dose of opioid administered in the PACU and floor including the background analgesia (PCA) and boluses. All opioids will be converted into mg intravenous (IV) morphine equivalent to standardize opioid consumption .
Time Frame: Initial 72 hours after surgery or until discharge, whatever comes first.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Gabapentin Enacarbil | Placebo
Number analyzed (Participants) | 28 | 32
mg | 4.0 (1.6) | 4.1 (1.7)
Statistical Analysis 1: Comparison: Gabapentin Enacarbil vs Placebo; Comparisons of opioid consumption were conducted independently for each study site. This analysis is for patients at the Cleveland Clinic main campus; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.77, Regression, Linear; Ratio of geometric means = 2.12, 95% CI 2-sided [0.21 to 18.54]
Statistical Analysis 2: Comparison: Gabapentin Enacarbil vs Placebo; Comparisons of opioid consumption were conducted independently for each study site. This analysis is for patients at the Cleveland Clinic Fairview hospital; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.09, Regression, Linear; Ratio of geometric means = 0.32, 95% CI 2-sided [0.03 to 3.16]

3. Secondary Outcome: Number of Participants With Persistent Pain 90-day After Surgery
Description: Number of participants with persistent pain at 90 days after surgery
Time Frame: within 90 days after surgery
Population: There were 5 participants in gabapentin enacarbil group and 4 in placebo group with missing value in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Enacarbil | Placebo
Number analyzed (Participants) | 23 | 28
Participants | 7 | 3
Statistical Analysis 1: Comparison: Gabapentin Enacarbil vs Placebo; Test type: Superiority; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 3.5, 98.75% CI 2-sided [0.5 to 24.3]

4. Secondary Outcome: Postoperative Nausea and Vomiting (PONV) up to 72 Hours After Surgery
Description: Postoperative nausea and vomiting (PONV) were recorded daily by nurses.
Time Frame: Initial 72 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Enacarbil | Placebo
Number analyzed (Participants) | 28 | 32
Participants | 8 | 12
Statistical Analysis 1: Comparison: Gabapentin Enacarbil vs Placebo; Test type: Superiority; p = 0.60, Regression, Logistic; Odds Ratio (OR) = 0.7, 98.75% CI 2-sided [0.2 to 3.1]

5. Secondary Outcome: Length of Hospital Stay in Hours
Description: Duration of hospitalization (hours) was recorded from the end of surgery to discharge, and compared between groups on the medians.
Time Frame: From the end of surgery to discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Gabapentin Enacarbil | Placebo
Number analyzed (Participants) | 28 | 32
hours | 78 [49 to 102] | 76 [56 to 82]

6. Secondary Outcome: Quality of Recovery (QoR-15) Score 72 Hours After Surgery
Description: Quality of Recovery (QoR-15) survey was assessed by blinded investigators at 72 hours after surgery or shortly before hospital discharge, whichever came first. It is a patient-reported outcome ranging from 0 to 150. The higher scale indicates better recovery.
Time Frame: Initial 72 hours after surgery or shortly before hospital discharge.
Population: There were 3 participants in gabapentin enacarbil group and 1 in placebo group with missing value in this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin Enacarbil | Placebo
Number analyzed (Participants) | 25 | 31
score on a scale | 114 (19) | 118 (15)

ADVERSE EVENTS:
Time Frame: Initial 72 hours after surgery or until hospital discharge, whichever came first.
Arm/Group | Gabapentin Enacarbil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 0/28 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT02840240/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT02840240/ICF_001.pdf